CLINICAL TRIAL: NCT06761664
Title: Decreasing Edema with Platysma Exercises Following Third Molar Extraction Surgery: a Randomized Controlled Trial
Brief Title: Decreasing Edema with Platysma Exercises Following Third Molar Extraction Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melek Volkan Yazici (Other)
Collaborators: Gazi University (Other); Ankara University (Other)
Responsible Party: Sponsor-Investigator, Melek Volkan Yazici, Assoc Prof., Yuksek Ihtisas University
Organization: Yuksek Ihtisas University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Platysma
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Third Molar Extraction
Keywords: Third molar extraction; Platysma muscle; Exercise; Edema
MeSH Terms: conditions — Motor Activity; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants in this group will perform exercises of the platysma muscle after third molar extraction surgery.
  Interventions: Other: Platysma Exercise Group
- Control (Usual treatment) (Active Comparator): Participants in this group will undergo routine treatment after third molar extraction surgery.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Other: Platysma Exercise Group — The participants in this group will perform a platysma exercise for 7 days following third molar extraction surgery.
  Arms: Intervention
Other: Control (Standard treatment) — Participants in this group will receive routine treatment following third molar extraction.
  Arms: Control (Usual treatment)

SUMMARY:
This study will investigate the effects of a platysma muscle exercise on edema following third molar extraction surgery.

DETAILED DESCRIPTION:
The investigators hypothesized that, during the muscle contraction of the platysma, the vascular structures will be subjected to a pump effect, leading to an increase in venous circulation. Additionally, due to its connection to the fascia, the investigators propose that platysma contractions may mobilize the fascia and stimulate the lymph nodes, thereby improving interstitial fluid flow. This could lead to an effective treatment option for decreasing edema after third molar tooth extraction. Therefore, this study aims to investigate the effects of platysma exercises applied after third molar tooth extraction on edema while observing the differences on pain and trismus.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-40,
* Those requiring impacted third molar extraction
* Those with no systemic health conditions, were included in the study
* Those who accepted to participate in the study

Exclusion Criteria:

* Those who had systemic diseases
* Those who were taking medications that could interfere with inflammation, or healing,
* Those who were pregnant or breastfeeding,
* Those who had infections or pathologies involving teeth 38 and 48,
* Those who were unable to comply with postoperative recommendations or required therapeutic interventions outside the study protocol

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Facial Edema | Change of facial edema from baseline to 7 days
  Edema will be measured by taking five distinct facial measurements using a standard plastic tape measure (accuracy ±0.5 mm), ensuring the tape makes contact with the skin. The following measurements will be recorded: (a) the distance between the most posterior point of the tragus and the most lateral point of the lip commissure; (b) from the tragus to the chin mid point; (c) from the tragus to the lateral canthus of the eye; (d) from the lateral canthus to the lowest point of the mandibular angle; and (e) from the mandibular angle to the middle of the nasal bone.

SECONDARY OUTCOMES:
Pain following third molar extraction | Change in pain scores from baseline to 7 days
  Pain will be assessed using a 100 mm visual analog scale. Patients will be asked to mark the point on the scale that best represented their level of pain. The scale ranges from 0, indicating no pain, to 10, representing the worst pain imaginable pain.
Trismus | Change of trismus from baseline to 7 days
  Trismus will be assessed by measuring the maximum inter-incisal distance using callipers to record the widest mouth opening.

CONTACTS AND LOCATIONS:
Overall Officials: GOKHAN YAZICI, A/Prof, Principal Investigator — Gazi University
Locations (1):
- Ankara University, Faculty of Dentistry, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to ethical reasons data can not be directly shared. Data can be provided upon request.